CLINICAL TRIAL: NCT06820528
Title: Trapeziectomy and Suture Suspensionplasty for Thumb Carpometacarpal Arthritis - Is In-Clinic Therapy Needed?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Nuelle (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Julie Nuelle, Assistant Professor, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-02062
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: CMC Arthritis; Occupational Therapy; Hand Arthritis
Keywords: CMC Arthroplasty; Thumb Arthritis; Hand Therapy
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be prospectively enrolled into two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occupational Therapy (Experimental): Participants in this arm will receive weekly occupational therapy for 6 weeks
  Interventions: Behavioral: Occupational Therapy
- Home Exercise (Active Comparator): Participants in this arm will complete an informal home exercise program provided by their treating physician
  Interventions: Behavioral: Home Exercise Program

INTERVENTIONS:
Behavioral: Occupational Therapy — Formal therapy with a certified hand therapist, weekly for 6 weeks
  Arms: Occupational Therapy
Behavioral: Home Exercise Program — A booklet on hand exercises to complete following surgery, including range of motion and strengthening exercises
  Arms: Home Exercise

SUMMARY:
The study is a randomized, controlled trial to evaluate the efficacy of formal occupational therapy on outcomes following CMC arthroplasty

DETAILED DESCRIPTION:
While hand surgeons agree that strength and flexibility exercises are crucial after surgery, there is currently no consensus on whether the benefits of participating in formal hand therapy outweigh the investment required. The financial and time investments required to participate in formal hand therapy can be particularly large in patients living in rural locations, as access to certified hand therapists are often limited. Therefore, a prospective, randomized trial of hand therapy utilization is warranted to explore this phenomenon. The purpose of this clinical trial is to assess the outcomes for post-operative therapy from in-clinic or at-home exercise therapies and analyze costs associated with the different therapies. For this clinical trial patients will be randomized to either in-clinic occupational therapy where patients come into clinic and undergo about 30-60 minutes of occupational therapy 1-2 a week with a physician or at-home exercise therapy where patients are provided instructions in clinic prior to HEP-therapy and have check-ins with physicians at their normal follow-up appointments; each consisting of about 5-10 minutes of exercise at home everyday of the week.

This study is a prospective, randomized, controlled trial to asses and analyze:

1. The outcomes after trapeziectomy and suture suspensionplasty with in-clinic occupational therapy (OT) and without in-clinic occupational therapy: home exercise program (HEP).
2. The cost difference between the OT and HEP groups as well as historical control patients that have undergone LRTI for thumb carpometacarpal joint arthritis (Including preoperative, intra-operative, and postoperative costs).

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years
* Patients undergoing CMC Arthroplasty
* Ability to read and write in English
* Ability to provide informed consent

Exclusion Criteria:

* Patients undergoing revision CMC arthroplasty
* Acute traumatic dislocation of the CMC joint as indication for surgery
* Concomitant treatment of MCP hyperextension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Kapandji Score | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  The Kapandji score is a widely used clinical metric for evaluating thumb opposition. It assesses the movement and functional reach of the thumb across into the palm and to the bases of the other fingers. The score ranges from 0 to 10, with each point representing the thumb's ability to touch distinct anatomical landmarks on the hand: from the radial side of the index finger base (score of 1) to the ulnar side of the little finger base (score of 10). This score helps in determining the functional impairment and potential recovery in cases involving thumb or hand injuries, often used in pre- and post-operative assessments.

SECONDARY OUTCOMES:
Radial Abduction (degrees) | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  Radial abduction refers to the movement of the thumb away from the hand's plane towards the radius, or the lateral side of the forearm. This motion is crucial for grasping larger objects and is an important aspect of hand function. It is commonly measured during hand and thumb functional assessments to evaluate the range of motion and strength, particularly after injury or surgery. Radial abduction is facilitated by several muscles, including the abductor pollicis longus, which plays a pivotal role in thumb movement and positioning.
Key Pinch Strength (kg) | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  Key pinch, also known as lateral pinch, involves the force applied between the thumb pad and the lateral side of the index finger. This specific type of pinch is crucial for activities that require precision, such as holding a key or grasping small objects. The key pinch is commonly assessed in occupational therapy and rehabilitation settings to evaluate hand function and grip strength, particularly after injury or in conditions affecting the nerves or muscles of the hand. Measurements are typically taken using a pinch gauge, which provides a quantitative value of pinch strength, helping in the assessment and monitoring of recovery progress.
Grip Strength (kg) | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  Grip strength is the force applied by the hand to pull or suspend objects and is a key indicator of hand function and overall health. It's measured using a dynamometer, an instrument that the individual squeezes with maximum effort.
PROMIS Upper Extremity | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Upper Extremity measure is a tool designed to assess self-reported upper extremity function. This measure evaluates the physical functioning and capability of the arms, shoulders, and hands based on the patient's perspective. Scores from this assessment are converted to a T-score metric, where 50 represents the mean of a relevant reference population, and each 10-point deviation represents one standard deviation from that mean. This standardization allows for the comparison of patient scores against population norms, which can be particularly useful in clinical trials, patient care, and research studies involving musculoskeletal health and rehabilitation.
PROMIS 29 | 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year
  The PROMIS-29 profile is a comprehensive tool that measures health across multiple domains using patient-reported outcomes. It evaluates seven key health domains along with pain intensity, offering a broad overview of a patient's health status. The domains include physical function, which assesses the ability to carry out physical activities; anxiety, evaluating feelings like fear and unease; depression, measuring feelings such as sadness and lack of interest; fatigue, assessing how often a patient feels tired; sleep disturbance, measuring perceptions of sleep quality; social roles and activities, evaluating the extent to which health limits participation in various activities; and pain interference, which assesses how pain hampers engagement in daily activities. Additionally, pain intensity is captured on a scale from 0 (no pain) to 10 (worst imaginable pain). Each domain consists of four questions, totaling 29 items. This tool is designed to be generic, suitable for a wide range of

CONTACTS AND LOCATIONS:
Overall Officials: Julia A.V. Nuelle, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data collected in this study, including potentially identifiable health information, we have decided not to share individual participant data with other researchers. This decision is guided by the need to strictly adhere to the privacy and confidentiality assurances provided to our participants at the time of consent. Moreover, the specific terms of participant consent do not allow for the sharing of their data beyond the scope of this research project.

REFERENCES:
- [Background] Stepan JG, Rolf L, Zhu E, Brody M, Landau AJ, Calfee RP, Dy CJ. Patient Perspectives after Trapeziectomy and Ligament Reconstruction Tendon Interposition: A Qualitative Analysis. Plast Reconstr Surg. 2022 Dec 1;150(6):1275e-1282e. doi: 10.1097/PRS.0000000000009676. Epub 2022 Sep 20. PMID 36126197
- [Background] Stirton JB, Kagy KL, Mooney ML, Jain MK, Skie M. Early Mobilization After Basal Joint Arthroplasty: Clinical Results. Hand (N Y). 2023 Mar;18(2_suppl):81S-86S. doi: 10.1177/15589447211038699. Epub 2022 Jan 26. PMID 35081799
- [Background] Hutchinson DT, Sueoka S, Wang AA, Tyser AR, Papi-Baker K, Kazmers NH. A Prospective, Randomized Trial of Mobilization Protocols Following Ligament Reconstruction and Tendon Interposition. J Bone Joint Surg Am. 2018 Aug 1;100(15):1275-1280. doi: 10.2106/JBJS.17.01157. PMID 30063589
- [Background] Barret PC, Hackley DT, Lockhart ES, Yu-Shan AA, Bravo CJ, Apel PJ. What Factors Influence Variability in Thumb Carpometacarpal Arthroplasty Care? A Survey of ASSH Members. Hand (N Y). 2025 Jan;20(1):129-135. doi: 10.1177/15589447231188454. Epub 2023 Aug 14. PMID 37575026
- [Background] Barrett PC, Hackley DT, Yu-Shan AA, Shumate TG, Larson KG, Deneault CR, Bravo CJ, Peterman NJ, Apel PJ. Provision of a Home-Based Video-Assisted Therapy Program Is Noninferior to In-Person Hand Therapy After Thumb Carpometacarpal Arthroplasty. J Bone Joint Surg Am. 2024 Apr 17;106(8):674-680. doi: 10.2106/JBJS.23.00597. Epub 2024 Apr 12. PMID 38608035